CLINICAL TRIAL: NCT02470507
Title: Evaluation of Immune Function in Patients With Acute Kidney Injury
Brief Title: Immune Function in Acute Kidney Injury
Status: Active, not recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: CSP88220
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- AKI with SIRS: Patients with AKI stage II or III and systemic inflammation without sepsis
  Interventions: Other: AKI
- AKI without SIRS: Patients with AKI stage II or III and no systemic inflammation
  Interventions: Other: AKI
- SIRS without AKI: Patients with systemic inflammation and normal renal function
  Interventions: Other: AKI
- No SIRS and no AKI: Patients after major surgery who do not have an infection, SIRS or AKI
  Interventions: Other: AKI

INTERVENTIONS:
Other: AKI — development of immune dysregulation and rise in inflammatory markers and activation of immune cells

SUMMARY:
The immune response to kidney damage during acute kidney injury (AKI) is an important contributor to the prolonged lack of renal function and progression of kidney injury. Most data related to intrarenal and interorgan pathways in AKI stem from animal research with sometimes conflicting results. Accurate evaluation of these processes in humans and identification of early diagnostic tools are critical for the development of strategies to prevent and attenuate AKI-related morbidity and mortality in patients.

The aim of this study is to evaluate immune function and miRNA expression in hospitalised patients with and without AKI.

DETAILED DESCRIPTION:
Hypothesis:

An overriding pro-inflammatory immune response underlies AKI in humans which contributes to dysfunction of non-renal organs

Principal research question:

Is AKI in humans associated with a predominantly pro-inflammatory immune response?

Secondary research questions:

1. Does AKI affect the phenotypic characterisation and function of neutrophils?
2. Does severity of AKI lead to differences in phenotypic characterisation and function of neutrophils?
3. What are the differences in cytokine profiles between AKI patients with and without systemic inflammation?
4. What are the differences in cytokine profiles between AKI patients with systemic inflammation and patients with systemic inflammation without AKI?
5. Is there a correlation between microRNA levels in patients with AKI and degree of AKI, renal recovery and patient outcome?

Study design:

Observational non-interventional study

Study population:

30 patients with AKI stage II or III * and systemic inflammation without sepsis 30 patients with AKI stage II or III * and no systemic inflammation 30 patients with systemic inflammation and normal renal function 30 patients after major surgery who do not have an infection, SIRS or AKI

* AKI will be defined by the KDIGO criteria

Primary outcome Detection of measurable phenotypic characteristics and function of leukocytes that are specific of patients with AKI.

Secondary outcomes:

1. Differences in phenotypic characterisation and function of neutrophils between patients with AKI stage II and III.
2. Differences in phenotypic characterisation and function of neutrophils between patients with and without AKI.
3. Differences in cytokine profiles between patients with AKI and systemic inflammation and patients with AKI without systemic inflammation
4. Differences in cytokine profiles between AKI patients with systemic inflammation and patients with systemic inflammation without AKI
5. Correlation between microRNA levels in patients with AKI and renal recovery
6. Correlation between microRNA levels in patients with AKI and patient outcome
7. Differences in cytokine profiles between AKI patients without systemic inflammation and patients without AKI and without systemic inflammation / infection.

Statistical analysis:

For the analysis of laboratory variables that describe the immunological phenotype, standard statistical methods will be applied. 1) When the normal distribution assumption is met, groups will be compared using ANOVA and the corresponding contrasts for group by group comparisons; 2) In the absence of normality or for ordinal variables, Kruskal Wallis will be applied for multi-group comparisons, and Wilcoxon for two-groups analysis. We will apply multiple testing correction via Benjamini-Hochberg FDR control.

For the analysis of miRNA array data, we will first follow the protocol quality control measures appropriate for the platform of choice, and subsequently will carry out statistical analysis using the SAMr and LIMMA packages from Bioconductor, via the R software. Similarly, for the analysis of PCR data, the package HTqPCR from bioconductor will be used for quality control. Depending on the distribution of the final data, either non-parametric statistics, or a moderated t-test will be applied for statistical comparisons, with the corresponding multiple testing corrections as above.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) admitted to the hospital (incl ICU) with one of the following:

  1. postoperative AKI II or III and systemic inflammation without sepsis
  2. systemic inflammation and normal renal function
  3. AKI II or III without systemic inflammation
  4. post-surgery with normal renal function and without SIRS or an infection

Exclusion Criteria:

* Renal transplant patients
* Patients on immunosuppressive drugs (except steroids)
* Patients with haematological malignancy
* Jehovah's witness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Phenotypic characteristics and function of leukocytes | 7 days

SECONDARY OUTCOMES:
Differences in phenotypic characterisation and function of neutrophils between AKI stage II and III. | 7 days
Differences in phenotypic characterisation and function of neutrophils between AKI and no AKI | 7 days
Differences in cytokine profiles between AKI + SIRS and AKI without SIRS | 7 days
Differences in cytokine profiles between SIRS + AKI and SIRS without AKI | 7 days
Correlation between microRNA levels in patients with AKI and renal recovery | 7 days
  Correlation between microRNA levels in patients with AKI and patient outcome Differences in cytokine profiles between AKI patients without systemic inflammation and patients without AKI and without systemic inflammation / infection.
Correlation between microRNA levels in patients with AKI and patient outcome | 7 days
  Differences in cytokine profiles between AKI patients without systemic inflammation and patients without AKI and without systemic inflammation / infection.
Differences in cytokine profiles between AKI patients without SIRS and patients without AKI and without SIRS | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas Foundation Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weller S, Varrier M, Ostermann M. Lymphocyte Function in Human Acute Kidney Injury. Nephron. 2017;137(4):287-293. doi: 10.1159/000478538. Epub 2017 Jun 30. PMID 28662513